CLINICAL TRIAL: NCT01014052
Title: Phase 1b Study to Evaluate QLT091001 in Subjects With Leber Congenital Amaurosis (LCA) or Retinitis Pigmentosa (RP) Due to Inherited Deficiencies of Retinal Pigment Epithelial 65 Protein (RPE65) or Lecithin:Retinol Acyltransferase (LRAT)
Brief Title: Safety/Proof of Concept Study of Oral QLT091001 in Subjects With Leber Congenital Amaurosis (LCA) or Retinitis Pigmentosa (RP) Due to Retinal Pigment Epithelial 65 Protein (RPE65) or Lecithin:Retinol Acyltransferase (LRAT) Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RET IRD 01
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: LCA (Leber Congenital Amaurosis); RP (Retinitis Pigmentosa)
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa | interventions — retinol acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: QLT091001 — oral QLT091001 administered once daily for 7 days

SUMMARY:
The purpose of this study is:

* to evaluate the safety of oral QLT091001
* to evaluate whether 7-day treatment with oral QLT091001 can improve visual function in subjects with LCA or RP due to RPE65 or LRAT mutations
* to evaluate duration of visual function improvement (if observed)

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with LCA or RP (with a mutation in either RPE65 or LRAT)

  * Subjects with LCA must be 5-65 years of age
  * Subjects with RP must be 18-65 years of age
* Subjects who have a "best-corrected" visual acuity of 3 letters or better (20/800 Snellen equivalent) or viable photoreceptors on OCT/FAF.

Exclusion Criteria:

* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 60 days of Day 0.
* Subjects with any clinically important abnormal physical finding at Screening.
* Subjects who have taken any prescription or investigational oral retinoid medication (e.g., Accutane,® Soriatane®) within 6 months of Day 0 and subjects who did not tolerate their previous oral retinoid medication will be excluded regardless of the time of last exposure.
* Subjects with a history of diabetes or chronic hyperlipidemia, hepatitis, pancreatitis, or cirrhosis.
* Subjects who have taken any supplements containing ≥10,000 IU vitamin A within 60 days of screening

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Visual Field | 12 months

SECONDARY OUTCOMES:
Vital signs, clinical laboratory tests, electrocardiogram (ECG), and adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sushanta Mallick, Study Director — QLT Inc.
Locations (7):
- United States (3):
  - The Chicago Lighthouse for People Who Are Blind or Visually Impaired (The Pangere Center For Inherited Retinal Diseases), Chicago, Illinois
  - Wilmer Eye Institute (Johns Hopkins University), Baltimore, Maryland
  - Scheie Eye Institute, Philadelphia, Pennsylvania
- Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec, Canada
- Institute for Ophthalmic Research, University of Tubingen, Tübingen, Germany
- The Rotterdam Eye Hospital, Rotterdam, Netherlands
- Moorefield Eye Hospital, London, United Kingdom

REFERENCES:
- [Derived] Scholl HP, Moore AT, Koenekoop RK, Wen Y, Fishman GA, van den Born LI, Bittner A, Bowles K, Fletcher EC, Collison FT, Dagnelie G, Degli Eposti S, Michaelides M, Saperstein DA, Schuchard RA, Barnes C, Zein W, Zobor D, Birch DG, Mendola JD, Zrenner E; RET IRD 01 Study Group. Safety and Proof-of-Concept Study of Oral QLT091001 in Retinitis Pigmentosa Due to Inherited Deficiencies of Retinal Pigment Epithelial 65 Protein (RPE65) or Lecithin:Retinol Acyltransferase (LRAT). PLoS One. 2015 Dec 10;10(12):e0143846. doi: 10.1371/journal.pone.0143846. eCollection 2015. PMID 26656277
- [Derived] Wen Y, Birch DG. Outer Segment Thickness Predicts Visual Field Response to QLT091001 in Patients with RPE65 or LRAT Mutations. Transl Vis Sci Technol. 2015 Oct 1;4(5):8. doi: 10.1167/tvst.4.5.8. eCollection 2015 Oct. PMID 26448901
- [Derived] Koenekoop RK, Sui R, Sallum J, van den Born LI, Ajlan R, Khan A, den Hollander AI, Cremers FP, Mendola JD, Bittner AK, Dagnelie G, Schuchard RA, Saperstein DA. Oral 9-cis retinoid for childhood blindness due to Leber congenital amaurosis caused by RPE65 or LRAT mutations: an open-label phase 1b trial. Lancet. 2014 Oct 25;384(9953):1513-20. doi: 10.1016/S0140-6736(14)60153-7. Epub 2014 Jul 13. PMID 25030840